CLINICAL TRIAL: NCT00775359
Title: Comparative, Randomized, Single-Dose, 2-Way Crossover Relative Bioavailability Study of Ranbaxy and Abbott (TriCor®) 160 mg Fenofibrate Tablets in Healthy Adult Volunteers Under Fed Conditions
Brief Title: Bioequivalence Study of Fenofibrate 160mg Tablets Under Fed Conditions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Ranbaxy Laboratories Limited (Industry)
Responsible Party: Dr. Tausif Monif, Ranbaxy Research Laboratories
Organization: Ranbaxy Inc. (Industry)
Allocation: Randomized | Model: Crossover | Masking: None
Other Study IDs: AA01824
Record Dates: First submitted 2008-10-17; First posted 2008-10-20 (Estimated); Last update posted 2008-10-20 (Estimated); Status verified 2008-10

CONDITIONS: Healthy
Keywords: bioequivalence fenofibrate tablets
MeSH Terms: interventions — Fenofibrate

STUDY DESIGN:
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- 1 (Experimental): Fenofibrate 160mg Tablets of Ranbaxy
  Interventions: Drug: Fenofibrate 160 mg tablets
- 2 (Active Comparator): TriCor® 160 mg Fenofibrate Tablets
  Interventions: Drug: Fenofibrate 160 mg tablets

INTERVENTIONS:
Drug: Fenofibrate 160 mg tablets

SUMMARY:
The objective of this study was to compare the single-dose relative bioavailability of Ranbaxy and Abbott (TriCor) 160 mg fenofibrate tablets under fed conditions.

DETAILED DESCRIPTION:
This was an open-label, randomized, single-dose, 2-way crossover, relative bioavailability study performed on 24 healthy adult male and female volunteers A total of 23 subjects (16 males and 7 females) completed the clinical phase of the study. In each period, subjects were housed from the evening before dosing until after the 24-hour blood draw. Subjects returned for all subsequent blood draws. Doses were separated by a washout period of 10 days.

Of the 24 healthy adult male and female volunteers enrolled in the study, 23 subjects (16 males and 7 females) completed the clinical phase of the study. Subject No. 10 failed to return for Period 2 check-in.

ELIGIBILITY:
Inclusion Criteria:

Subject candidates must fulfill the following inclusion criteria to be eligible for participation in the study, unless otherwise specified:

* Healthy adult male and female volunteers, 18-55 years of age;
* Weighing at least 52 kg for males and 45 kg for females and within 15% of their ideal weights (Table of "Desirable Weights of Adults", Metropolitan Life Insurance Company, 1983);
* Medically healthy subjects with no clinically abnormal laboratories and ECGs, as deemed by the principal investigator;
* Females of childbearing potential should either be sexually inactive (abstinent) for 14 days prior to the study and throughout the study or be using one of the following acceptable birth control methods:

  * Surgically sterile (tubal ligation, hysterectomy, bilateral oophorectomy) 6 months minimum. Proof is required for the hysterectomy and oophorectomy;
  * IUD in place for at least 3 months;
  * Barrier methods with spermicide (condom, diaphragm) for at least 14 days prior to the start of the study and throughout the study;
  * Surgical sterilization of the partner (vasectomy for 6 months minimum);
  * Hormonal contraceptives for at least 3 months prior to the start of the study. Other birth control methods may be deemed acceptable.
* Postmenopausal women with amenorrhea for at least 2 years;
* Voluntary consent to participate in the study.

Exclusion Criteria:

Subject candidates must not be enrolled in the study if they meet any of the following criteria:

* History or presence of significant: cardiovascular, pulmonary, hepatic, renal, hematologic, gastrointestinal, endocrine, immunologic, dermatologic, neurologic or psychiatric disease.
* In addition, history or presence of:

  * alcoholism or drug abuse within the past 2 years;
  * hypersensitivity or idiosyncratic reaction to fenofibrate or other lipid regulating agents.
* Female subjects who are pregnant or lactating.
* Subjects who have been on an abnormal diet (for whatever reason) during the 30 days prior to the first dosing.
* Subjects who have made a donation (standard donation amount or more) of blood or blood products (with the exception of plasma as noted below) within 30 days prior to the study.
* Subjects who have made a plasma donation within 7 days prior to the study.
* Subjects who have participated in another clinical trial within 30 days prior to the first dose.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 24 (Actual)
Dates: Start 2002-08; Primary Completion 2002-09 (Actual); Study Completion 2002-10 (Actual)

PRIMARY OUTCOMES:
Bioequivalence

CONTACTS AND LOCATIONS:
Locations (1):
- MDS Pharma Services, Phoenix, Arizona, United States

REFERENCES:
- See also: Related Info — http://clinicalstudies.ranbaxy.com
- See also: Related Info — http://dailymed.nlm.nih.gov/dailymed/about.cfm
- See also: Related Info — http://www.fda.gov/opacom/7alerts.html